CLINICAL TRIAL: NCT01673373
Title: ARTISAN: iCAST™ RX De Novo Stent Placement for the Treatment of Atherosclerotic Renal Artery Stenosis in Patients With Resistant Hypertension
Brief Title: Renal Stent Placement for the Treatment of Renal Artery Stenosis in Patients With Resistant Hypertension
Acronym: ARTISAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atrium Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iCAST™ RX-ARAS-001
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Renal Artery Stenosis; Hypertension, Renovascular
Keywords: Renal Artery Stenosis; Renal Artery Obstruction; Renovascular Hypertension; Resistant Hypertension; Renal Revascularization; Atherosclerotic Renal Artery Stenosis; Atherosclerotic Renal Artery Stenosis (ARAS); Renal Artery Stenosis (RAS); Uncontrolled hypertension; Hypertension; Systolic blood pressure; Blood pressure
MeSH Terms: conditions — Renal Artery Obstruction; Hypertension, Renovascular; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- iCAST RX™ Stent Systen (Experimental): All enrolled subjects will receive the iCAST RX™ Stent System
  Interventions: Device: iCAST™ Rx Stent System

INTERVENTIONS:
Device: iCAST™ Rx Stent System — All enrolled subjects will undergo primary stenting of the target lesion(s) by placement of the iCAST™ RX Stent System.
  Other Names: iCAST™ RX

SUMMARY:
The purpose of this trial is to test how well the iCAST™ RX Stent works in patients diagnosed with atherosclerotic renal artery stenosis and whether or not increased blood flow by the stent will help to control blood pressure.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multicenter clinical trial that will take place at up to 25 US/ Outside US (OUS) sites. Primary endpoints have been determined to show the safety, effectiveness, and clinical outcomes of the iCAST™ RX Stent System. Safety and effectiveness will be evaluated based on the primary patency rate at 9-months on a per lesion basis evaluated against a performance goal of published studies with bare-metal stents. The primary clinical endpoint will assess the improvement in Systolic Blood Pressure (SBP) at 9-months as compared to baseline Systolic Blood Pressure.

Eligible subjects will undergo a two-week Medical Documentation Screening period to confirm resistant hypertension (SBP ≥ 155mmHg) while on maximum tolerable doses of ≥ three anti-hypertensive medications from at least three distinct classes of drugs, one of which must be a diuretic.

There must be documented clinical evidence to support likelihood of angiographic findings > 80% whether it is Duplex Ultrasound (DUS), Computed Tomography angiogram (CTa), Magnetic Resonance angiogram (MRa) or other medical evidence. After meeting screening and clinical eligibility criteria, subjects will undergo a baseline assessment for angiographic eligibility. After angiographic documentation of a ≥ 80% renal artery stenosis or Fraction Flow Reserve (FFR) < 0.8 is confirmed, the subject may be enrolled in the trial by placement of the investigational device.

The 9-month visit will include a follow-up DUS of the target renal artery. If the DUS is non-diagnostic due to an imaging problem, such as overlying bowel gas or body habitus, a second DUS may be attempted. If the DUS is indicative of ≥ 60% stenosis as determined by the core laboratory, or the second DUS remains non-diagnostic, a contrast angiogram will be used to assess the degree of restenosis of the covered stent(s).

Clinical follow-up visits will be required for all enrolled subjects at 30-days, 9-months, 12-months, 24-months, and 36-months. A 6-month and 18-month visit will occur via telephone to collect medication usage and Adverse Events (AEs) only. The 36-month clinic office visit will be required as the final safety visit.

ELIGIBILITY:
General Inclusion Criteria:

1. Age ≥ 18 at the time of informed consent.
2. Subject or subject's legal representative have been informed of the nature of the trial, agrees to participate, and has signed an Institutional Review Board (IRB)/Ethics Committee (EC) approved Informed Consent Form (ICF).
3. Subjects that have bilateral kidneys or a solitary functioning kidney with Renal Artery Stenosis in at least one kidney and an average Systolic Blood Pressure (SBP) ≥ 155mmHg.
4. Subject has a history of maximum tolerable dose of ≥ 3 anti-hypertensive medications of different classes, one of which must be a diuretic (for at least two weeks prior to Medical Documentation Screening period).

   a. A documented history for a minimum of 3 months showing reasonable and aggressive efforts to manage hypertension prior to consent. This must include the use of a broad variety of medications that have been used and failed or not tolerated.
5. Subject must have documented clinical evidence to support likelihood of angiographic findings > 80% whether it is DUS, CTa, MRa or other medical evidence.
6. New York Heart Association (NYHA) class I, II, or III the time of trial enrollment.

Note: When a subject has bilateral Renal Artery Stenosis both of which require stenting, it is recommended to treat both kidneys with an iCAST™ RX Stent System during the index procedure. In the event that a subject needs a renal stenting procedure staged for renal protection, it is important that the Investigator treats the second renal artery with an iCAST™ RX Stent System after 30 days of the index procedure. If subjects with bilateral stenosis have only one lesion that meets protocol inclusion criteria that lesion should be treated per protocol. The recommendation is to NOT treat the second non-qualifying lesion, however if the operator feels strongly it is indicated, then they should treat per standard of care after 30-days post index procedure in order to comply with exclusion criteria #10.

Subjects with flash pulmonary edema are allowed into the trial should they meet all other Inclusion and Exclusion criteria.

Angiographic Anatomic Inclusion Criteria:

1. Angiographic diameter renal artery stenosis ≥ 80% involving unilateral or bilateral renal arteries.

   a. The degree of percent diameter stenosis for all lesions intended to be treated, must be confirmed via one of the following methods: i. Manual or automated measurement with calipers ii. Measured Flow Fraction Reserve (FFR) < 0.8 using a pressure wire iii. Measured translesional peak pressure gradient of > 21 mmHg after induced hyperemia via dopamine or papaverine using a 4 Fr or less catheter or pressure wire.

   b. Subjects with 60-79% angiographic stenosis who have confirmed FFR < 0.8 may be enrolled.
2. Renal pole-to-pole length > 8cm (per visual estimate).
3. Target lesion length ≤ 16mm per vessel (per visual estimate).
4. Renal artery vessel diameter ≥ 5.0mm and ≤ 7.0mm (per visual estimate).
5. Lesion originating ≤ 15mm of the renal ostium.

General Exclusion Criteria:

1. Subject's estimated life expectancy is < 12 months.
2. Subject has a history of transplanted kidney(s), has had another recent organ transplant or polycystic kidney disease.
3. Subject with estimated glomerular filtration rate (eGFR) ≤ 25 mL/min/1.73 m2
4. Subject has a history of bleeding diathesis or coagulopathy or refuses blood transfusions.
5. Subject has a known contraindication to heparin, aspirin, thienopyridine, other anti-coagulant/antithrombotic therapies, contrast media, stainless steel, and/or polytetrafluoroethylene (PTFE).
6. Subject has had a previous renal bypass operation, a bypass is planned, or the target lesion is located within or beyond a bypass graft.
7. Subject has received a thrombolytic agent within the past 30 days.
8. Subject has documented acute pulmonary edema or systolic heart failure with ejection fraction < 30% and/or hospitalization requiring intubation and ventilation support for this diagnosis within the previous 90 days or hypertensive emergencies defined as resulting in organ damage.
9. Concurrent enrollment in any investigational trial wherein subject's participation has not been completed.
10. Subject has had a planned or anticipated cardiovascular surgical or interventional procedure outside of the affected renal artery (including, but not limited to, aortic, renal, cardiac, carotid, femoro-popliteal, and below the knee) within 30 days prior to the index procedure and prior to completion of the 30 day follow-up.
11. Subject has suffered a stroke or Transient Ischemic Attack (TIA) in the past 3 months.
12. Subject is pregnant, lactating, or is of child-bearing potential and plans to become pregnant during the follow-up trial period.
13. Subject with significant valvular disease.
14. Subject with known significant proteinuria > 2+ or > 2.0gm/d.
15. Subject with known bilateral upper-extremity arterial stenosis that result in spuriously low arm pressures or without the ability to gain reliable blood pressure measurements in at least one upper extremity.
16. Subject with active sepsis.
17. Subject with serum creatinine ≥ 3.0mg/dL.
18. Subject with NYHA Class IV at the time of enrollment.
19. Subject is on hemodialysis.
20. Subject has a history of renal aneurysm.
21. Subject with cardiogenic shock.
22. Subject with cardiomyopathy.
23. Subject has an uncontrolled concurrent illness, including but not limited to ongoing or active infection or active autoimmune disease requiring immunosuppressive therapy.
24. Any subject with clinically significant cardiovascular, respiratory, neurologic, hepatic, endocrine, major systematic disease, making implementation or interpretation of the protocol or protocol results difficult or who in the opinion of the investigator would not be a good candidate for enrollment.

Angiographic Anatomic Exclusion Criteria:

1. The planned site of intervention is totally occluded or has an anatomic configuration likely to prohibit adequate dilatation, and/or passage or implantation of the investigational device.
2. Subject has multiple ipsilateral lesions of the target renal artery that cannot be covered by a single stent.
3. There is a previously implanted stent in the target vessel or there is a previously implanted stent in the contralateral vessel < one year.
4. Subject has fibromuscular dysplasia, in renal artery and/or other vascular bed.
5. The target lesion site is associated with a thrombus.
6. Target lesion treated with laser atherectomy, directional atherectomy or other adjuncts to percutaneous balloon angioplasty (PTA).
7. Subject has a critical stenotic (> 70%) small accessory renal artery.
8. Subject has an abdominal aortic aneurysm > 4.0cm in diameter or a severe atherosclerotic aorta.
9. Main renal artery length ≤ 15mm precluding the safe deployment of a covered renal stent.
10. Any lesion that would include blocking of renal artery side branch.
11. Renal artery stenosis due to dissection of renal artery: spontaneous or traumatic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-10-23 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2020-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Rosenfield, MD, Principal Investigator — Massachusetts General Hospital; Gary Ansel, MD, Principal Investigator — OhioHealth Research Institute
Locations (12):
- United States (12):
  - Mission Cardiovascular Research Institute, Fremont, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Clearwater Cardiovascular and Interventional Consultants, Clearwater, Florida
  - Advocate Health and Hospitals Corporation, Naperville, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beaumont Health Systems, Royal Oak, Michigan
  - Holy Name Medical Center, Teaneck, New Jersey
  - Mid Carolina Cardiology, Charlotte, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - OhioHealth Research Institute, Columbus, Ohio
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Tennova Healthcare - Turkey Creek Medical Center, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- iCAST™ RX Stent System: All enrolled subjects, defined as patients that underwent primary stenting of the target lesion(s) by placement of the iCAST™ RX Stent System.
Period: Overall Study
Arm/Group | iCAST™ RX Stent System
Started | 68
Completed | 66 (Completed primary endpoint follow up.)
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | iCAST™ RX Stent System
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 53
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 68
Number of Qualifying Lesions [Count of Participants; unit: Participants]
  Unilateral | 54
  Bilateral | 14
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 166.2 (12.19)

OUTCOME MEASURES:

1. Primary Outcome: Primary Patency
Description: Primary patency rate at 9 months was defined as continuous patency without the occurrence of a total occlusion of the original lesion, without a re-intervention to treat a partial or total occlusion of the stented segment, or bypass of the stented segment due to clinically-driven restenosis or occlusion.
Time Frame: 9 months
Population: Subset of enrolled subjects with available duplex ultrasound or angiography assessment within the 9-month visit window.
Measure: Count of Units; unit: Subject-lesions
Units Other Than Participants: Subject-lesions
Arm/Group | iCAST™ RX Stent System
Number analyzed (Participants) | 56
Number analyzed (Subject-lesions) | 70
Subject-lesions | 66
Statistical Analysis 1: Comparison: iCAST™ RX Stent System; The original Performance Goal of 70% patency rate was derived from a thorough literature review of trials with renal bare metal stent placement. Other assumptions included a determination of samples size based upon a one-sided alpha of 0.025 and desired power of 87%, and assumption of 10% attrition. The null hypothesis was that the incidence of primary patency at 9 months is less than or equal to 70%; Test type: Other — Due to the early termination of enrollment, all inferential analyses were interpreted as descriptive and carried out in an exploratory manner; p < .0001, one-sided exact — The p-value was computed using a one-sided exact test of the difference between the observed rate and the Performance Goal (equal to 70%). The defined threshold for statistical significance is .025; The cumulative incidence of primary patency was computed as the number of subject-lesions with primary patency at 9 months divided by the number of subject-lesions and was analyzed using the allowable window of 243 to 303 trial days. An exact binomial one-sided 95% CI was constructed and the lower limit compared to the Performance Goal equal to 70%

2. Primary Outcome: Systolic Blood Pressure
Description: Change in systolic blood pressure (SBP) at 9 months as compared to baseline SBP.
Time Frame: Baseline and 9 months
Population: Subset of enrolled subjects with available blood pressure data at baseline and 9 months.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | iCAST™ RX Stent System
Number analyzed (Participants) | 63
mmHg | 15.7 (21.20)
Statistical Analysis 1: Comparison: iCAST™ RX Stent System; The primary endpoint of systolic blood pressure was analyzed according to the Performance Goal of a decrease in systolic blood pressure of 10 mmHg between procedure and 9 months; Test type: Other — A one-sided 95% Confidence Interval for the mean difference between baseline and 9-month systolic blood pressure was constructed and the lower limit compared to the 10 mmHg performance goal. A p-value of the difference between the estimated systolic blood pressure change from the baseline and the performance goal was computed using a paired t-test; p = .0192, t-test, 1 sided — The defined threshold for statistical significance is .025

3. Secondary Outcome: Procedure-Related Major Adverse Events (MAE)
Description: The occurence of procedure-related MAEs is reported as a percentage of subjects with MAE. Inclusive of:
  1. Procedure- or device-related occurrence of death
  2. Q-Wave myocardial infarction (MI)
  3. Clinically driven target lesion revascularization (TLR)
  4. Significant embolic events defined as unanticipated kidney/bowel infarct, clinically driven by symptoms of abdominal or back pain and confirmed with CT scan or open surgery; lower extremity ulceration or gangrene; or kidney failure.
Time Frame: 30 days, 9 months
Population: All enrolled subjects, defined as patients that underwent primary stenting of the target lesion(s) by placement of the iCAST™ RX Stent System.
Measure: Count of Participants; unit: Participants
Arm/Group | iCAST™ RX Stent System
Number analyzed (Participants) | 68
Participants
  Overall subjects experiencing MAE | 5
  MAE within 30 days | 0
  MAE within 9 months | 2

4. Secondary Outcome: Technical Success
Description: Technical success is defined as successful delivery and deployment of the iCAST™ RX Stent System with ≤ 30% residual angiographic stenosis after covered stent deployment (including post-dilatation) assessed via quantitative vascular analysis (QVA) by an independent core laboratory.
Time Frame: Day of Procedure
Population: All enrolled subjects, defined as patients that underwent primary stenting of the target lesion(s) by placement of the iCAST™ RX Stent System. Note that analysis is per subject lesion with available angiography.
Measure: Count of Units; unit: Subject-lesions
Units Other Than Participants: Subject-lesions
Arm/Group | iCAST™ RX Stent System
Number analyzed (Participants) | 68
Number analyzed (Subject-lesions) | 81
Subject-lesions | 81

5. Secondary Outcome: Acute Procedural Success
Description: Acute procedural success is defined as technical success without the occurrence of MAE prior to hospital discharge.
Time Frame: Day of Procedure, prior to hospital discharge
Population: as for outcome 4
Measure: Count of Units; unit: Subject-lesions
Units Other Than Participants: Subject-lesions
Arm/Group | iCAST™ RX Stent System
Number analyzed (Participants) | 68
Number analyzed (Subject-lesions) | 81
Subject-lesions | 81

6. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: Target Lesion Revascularization (TLR) is measured as the proportion of subjects-lesions that require a clinically-driven reintervention of the target lesion through 9 months.
  a. A clinically-driven TLR is defined as a TLR (percutaneous balloon angioplasty (PTA), bare metal stent or repeat covered stent deployment, or surgical bypass) due to documented recurrent hypertension from 30-days post-procedure level and/or deterioration in renal function from baseline value, associated with angiographic core laboratory adjudication of a ≥ 60% diameter covered stent restenosis.
Time Frame: 9 months
Population: All enrolled subjects, defined as patients that underwent primary stenting of the target lesion(s) by placement of the iCAST™ RX Stent System. Note that analysis is per subject lesion.
Measure: Count of Units; unit: Subject-lesions
Units Other Than Participants: Subject-lesions
Arm/Group | iCAST™ RX Stent System
Number analyzed (Participants) | 68
Number analyzed (Subject-lesions) | 82
Subject-lesions | 3

7. Secondary Outcome: Rate of Incidental TLR
Description: The rate of incidental TLR is the rate of TLRs not meeting the definition of a clinically-driven TLR.
Time Frame: 9 months
Population: as for outcome 6
Measure: Count of Units; unit: Subject-lesions
Units Other Than Participants: Subject-lesions
Arm/Group | iCAST™ RX Stent System
Number analyzed (Participants) | 68
Number analyzed (Subject-lesions) | 82
Subject-lesions | 2

8. Secondary Outcome: Systolic Blood Pressure (SBP) Control
Description: The change in SBP from baseline to 30 days
Time Frame: Baseline and 30 days
Population: Subset of enrolled subjects with available blood pressure measurements at both time points.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | iCAST™ RX Stent System
Number analyzed (Participants) | 67
mmHg | -13.6 (18.83)

9. Secondary Outcome: SBP Control
Description: The change in SBP from baseline to 9 months
Time Frame: Baseline and 9 months
Population: Subset of enrolled subjects with available blood pressure measurements at both time points.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | iCAST™ RX Stent System
Number analyzed (Participants) | 63
mmHg | -15.7 (21.20)

10. Secondary Outcome: Secondary Patency Rate
Description: Secondary patency rate at 9 months after a clinically-driven TLR which restores patency after total occlusion.
Time Frame: 9 months
Population: as for outcome 6
Measure: Count of Units; unit: Subject-lesions
Units Other Than Participants: Subject-lesions
Arm/Group | iCAST™ RX Stent System
Number analyzed (Participants) | 68
Number analyzed (Subject-lesions) | 82
Subject-lesions | 3

11. Secondary Outcome: Change in Number of Anti-Hypertensive Medications
Description: Change in number of anti-hypertensive medications as compared to baseline.
Time Frame: Baseline and 9 months
Population: Subset of enrolled subjects with available medication information.
Measure: Mean (Standard Deviation); unit: Number of Anti-hypertensive Medications
Arm/Group | iCAST™ RX Stent System
Number analyzed (Participants) | 63
Number of Anti-hypertensive Medications | -0.1 (0.76)

12. Secondary Outcome: Change in Renal Function
Description: Renal function compared to baseline as measured by estimated Glomerular Filtration Rate (eGFR) at 30 days.
Time Frame: Baseline and 30 days
Population: Subset of enrolled subjects with available eGFR measurements.
Measure: Mean (Standard Deviation); unit: eGFR mL/min/1.73 m^2
Arm/Group | iCAST™ RX Stent System
Number analyzed (Participants) | 67
eGFR mL/min/1.73 m^2 | -0.5520 (8.42795)

13. Secondary Outcome: Change in Renal Function
Description: Renal function compared to baseline as measured by estimated Glomerular Filtration Rate (eGFR) at 9 months.
Time Frame: Baseline and 9 months
Population: Subset of enrolled subjects with available eGFR measurements.
Measure: Mean (Standard Deviation); unit: eGFR mL/min/1.73 m^2
Arm/Group | iCAST™ RX Stent System
Number analyzed (Participants) | 65
eGFR mL/min/1.73 m^2 | -1.9964 (13.42781)

ADVERSE EVENTS:
Time Frame: Non-serious Adverse Events were reported through 9 months. Serious Adverse Events were reported through 3 years.
Description: Note that the adverse events reported are those reported through the cut off date related to the primary endpoint analysis.
Arm/Group | iCAST™ RX Stent System
All-Cause Mortality (participants affected / at risk) | 4/68
Serious Adverse Events (participants affected / at risk) | 40/68
Other Adverse Events (participants affected / at risk) | 12/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iCAST™ RX Stent System (N=68)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 7 (7)
Arrhythmia (Cardiac disorders) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 6 (6)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1)
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Device occlusion (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Urinary tract infection (Infections and infestations) | 2 (2)
Arterial restenosis (Injury, poisoning and procedural complications) | 8 (9)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 4 (4)
Depression (Psychiatric disorders) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Brachiocephalic artery occlusion (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 2 (2)
Intermittent claudication (Vascular disorders) | 2 (2)
Malignant hypertension (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 2 (2)
Subclavian artery aneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iCAST™ RX Stent System (N=68)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)

LIMITATIONS AND CAVEATS:
The limitation of the study was the termination of enrollment due to the change in clinical practice.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-07-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT01673373/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT01673373/SAP_001.pdf